CLINICAL TRIAL: NCT03049527
Title: Understanding Occupational and Non-occupational Risks Associated With CKDu in Sugarcane Workers in Guatemala
Brief Title: CKDu in Sugarcane Workers in Guatemala
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Pantaleon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 16-1824
Record Dates: First submitted 2017-01-31; First posted 2017-02-10 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Unknown Origin
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The single group will receive an intervention of enhanced education and incentives aimed at increasing hydration and reducing heat stress.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Education, Incentives and Feedback (Experimental): Education, Incentives and Feedback are all directed to all study participants.
  Interventions: Behavioral: Education, Incentives and Feedback

INTERVENTIONS:
Behavioral: Education, Incentives and Feedback — The study participants will receive additional educational activities, including low-literacy fact sheets on liquid intake guidelines, cards with instructions on how to self-monitor urine color and volume, and flyers and posters placed throughout the worksite. All consenting study participants will be offered incentives to start the work day hydrated and then to maintain or improve their hydration status over the work shift. Participants who do not meet hydration goals will receive additional coaching and feedback on ways to improve hydration.Feedback will also be provided to all groups about their productivity level to help participants recognize the connection between improved health and function.

SUMMARY:
The objective of this research project is to investigate specific behaviors and exposures related to sugarcane work and their association with non-communicable diseases, specifically Chronic Kidney Disease of Unknown Origin (CKDu) among sugarcane workers in Guatemala. Over the course of the 6-month sugarcane harvest the investigators will assess risk factors for declining kidney function, and also changes in biomarkers of kidney function pre and post work shift of field and factory workers and their possible relationships with dehydration and heat stress. The investigators will also evaluate the effectiveness of an intervention aimed at increasing hydration and reducing heat stress. Finally the investigators will measure biomarkers of exposure and environmental samples for heavy metals, agrochemicals, and infectious disease (Leptospira).

DETAILED DESCRIPTION:
This protocol describes two prospective cohort studies and one intervention study that will be conducted throughout the sugarcane harvest, from October through May, at Pantaleon's sugarcane plantations in Guatemala.

Overview of Studies

The investigators propose to conduct the three studies by making use of existing pre-employment data from prior years and by collecting new data during the 6-month sugarcane harvest. Pre-employment data are collected for all workers (N=5000) by Pantaleon and screenings occur throughout the harvest. Pre-employment and screening data include information on demographics, behaviors, work practices, non-communicable diseases, including kidney disease.

The purpose of the three new studies will be to collect detailed data on risk factors and biomarkers for CKDu. Risk factors will be assessed by collecting information through surveys and medical exams, and by collecting biological samples (blood and urine) from a subsample of the workers.

Study 1) Natural History of CKDu Study

Study Rationale: This study will prospectively follow a cohort of sugarcane workers (N=407) over multiple years to understand the natural history of CKDu. By following this cohort of workers, we will be able to describe the prevalence and incidence of abnormal eGFR and identify risk factors for CKDu.

Study Design and Populations: Pantaleon conducted a post-harvest evaluation of 407 workers following the 2015-2016 harvest. The investigators will conduct a prospective longitudinal study of this established cohort of workers (recruited during the end of the 2015-16 harvest) and will work with Pantaleon to replicate this post-harvest evaluation at the end of the 2016-2017 harvest.

Study 2) Industrial Mill Worker Observational Study

Study Rationale: This study will prospectively follow a stratified random selection of 100 mill workers throughout the harvest to understand the prevalence and incidence of kidney damage. The investigators will be able to describe the prevalence and incidence of abnormal eGFR and identify risk factors for CKDu. Although mill workers are indoors, we have informally observed that some of them work under conditions of high heat, placing them at risk for heat stress, dehydration and possibly CKDu.

Study Design and Population: Occupational Health and Safety staff at Pantaleon have identified job descriptions associated with heat exposure in the mill. Pantaleon will conduct pre-employment evaluations among 100 mill workers, specifically selecting a random sample of workers with job titles associated with high heat. At the end of the harvest, the investigators will collect occupational and non-occupational risk factors through a survey and medical exam and measure creatinine levels through a blood finger prick among the 100 mill workers.

Study 3) Hydration Study

Study Rationale: This study will prospectively assess acute and chronic kidney damage among sugarcane workers by evaluating kidney function a) before the start of the harvest and at the end of the harvest, and b) before and after work shifts during the harvest. An intervention will be implemented aimed at increasing hydration and reducing heat stress among sugarcane workers throughout the day. The investigators will assess the effectiveness of this intervention in increasing hydration and work productivity, with the final goal of the intervention aimed at decreasing acute and chronic kidney damage.

Study Design and Population: This study will comprise of the following: 1) implementation of an intervention which will include a wellness incentive and enhanced education on heat stress and hydration, and 2) investigation of biological markers of dehydration and acute kidney injury among approximately 500 sugarcane workers. Workers will be recruited from 10 work groups randomly selected at the Pantaleon work site. Each group will have data collected 3 times during the 6-month harvest.

Sub-Study 3.1) Heat Sub-study

Study Rational: This sub-study will increase understanding of the physiological response of workers to heat exposure and determine the workers' metabolic workload. The investigators will be able to examine across shift changes of physiological responses and its effects on acute and chronic kidney function. It will help determine if workers are receiving sufficient duration and number of rest periods.

Study Design and Population: Among the participants of the Hydration study, 100 workers will be randomly selected to participate in the Heat study. Data for this study will be collected during 3 periods of the Hydration Study (November, January, and March). When each Heat Sub-study participant is having data collected for the Hydration Study, the investigators will collect this additional information for that participant.

ELIGIBILITY:
Inclusion Criteria:

* currently employed by Pantaleon
* age 18 or older.

Exclusion Criteria:

* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 531 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
Change in Abnormal Glomerular Filtration Rate (eGFR) | Day 0 then every 4 weeks for 8 weeks
  Calculated from serum creatinine levels measured in blood samples. Abnormal eGFR is defined as an eGFR of <60 ml/min/1.73 m2. Serum creatinine will be used to calculate eGFR using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation for all participants. Lower eGFR and higher serum creatinine levels indicate worse kidney function.

SECONDARY OUTCOMES:
Change in Prevalence of Workplace Injuries and Illnesses | Week 1 and 6 months
  Self-reported injuries and illness will be collected via the surveys, which we will use to compare with data collected in the field by Pantaleon's health auxiliary nurses. All data collected will be de-identified as described in detail below. In addition, the incidence of non-communicable diseases will be examined in the Pantaleon study such as diabetes, hypertension, and obesity. Participants will be classified as having diabetes or hypertension if they reported a history of or were currently treated for diabetes or hypertension. Participants will be classified as obese if their body mass index was ≥30 kg/m2 (based on World Health Organization classifications). In addition, incidence of symptoms indicative of the infectious disease Leptospirosis will be collected.
Change in Productivity | Over the 6 month harvest period
  Reported from Pantaleon's daily records of tons of cane produced per worker.

CONTACTS AND LOCATIONS:
Overall Officials: Lee Newman, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States
- Panteleon, Escuintla, Guatemala

IPD SHARING:
Plan to Share IPD: No